CLINICAL TRIAL: NCT04681027
Title: A Multicenter Study of the Safety, Tolerability, Effectiveness, and Pharmacokinetics of Oxymorphone HCL Extended-Release Tablets in Pediatric Subjects Requiring an Around-The-Clock Opioid for an Extended Period of Time
Brief Title: Safety, Tolerability, Effectiveness, and Pharmacokinetic Data in Opioid-experienced Children
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Suspended 06Feb2020 per FDA Request
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN3202-037
Record Dates: First submitted 2020-12-03; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain; Postsurgical Pain
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative | interventions — Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pediatric Age Groups: 7 to ≤12 years (Active Comparator): Participants expected to require ATC opioids for an extended period of time
  Interventions: Drug: Oxymorphone hydrochloride (HCl)
- Pediatric Age Groups: 13 to ≤17 years (Active Comparator): Participants expected to require ATC opioids for an extended period of time
  Interventions: Drug: Oxymorphone hydrochloride (HCl)

INTERVENTIONS:
Drug: Oxymorphone hydrochloride (HCl) — Opioid
  Other Names: OPANA® ER (oxymorphone HCl) Extended-Release Tablets

SUMMARY:
The purpose of this study was to assess the safety and pharmacokinetics (single- and multiple-dose) of oxymorphone ER for the relief of moderate to severe pain in pediatric participants ages 7 - ≤17 years old requiring a continuous, around-the-clock (ATC) opioid treatment for an extended period.

ELIGIBILITY:
Inclusion Criteria:

1. Were males or females 7 - ≤17 years of age. Females of childbearing potential had to be practicing abstinence or using a medically acceptable form of contraception (eg, intrauterine device, hormonal birth control, or double barrier method). For the purpose of this study, all menstruating females were considered to be of childbearing potential unless they were biologically sterile or surgically sterile for more than 1 year.
2. Had chronic pain (malignant and/or nonmalignant) or postsurgical pain expected to require ATC opioid analgesia for up to 12 weeks with at least 10 mg per day oxymorphone ER (approximately equal to 30 mg per day oral MSE).
3. Had a body weight at least 18 kg.
4. Were able to swallow oxymorphone ER tablets.
5. Had laboratory results from within 21 days prior to Baseline available including clinical chemistry and hematology laboratory analytes. Intraoperative (prior to surgical incision) labs were acceptable provided the results had been reviewed by the investigator for study eligibility prior to dosing.
6. Subjects with postsurgical pain were prescribed a parenteral analgesic regimen utilizing a short-acting opioid analgesic AND were anticipated to be switched to an oral opioid for an extended period of time (according to institutions standard of care).
7. Were able to provide pain assessment evaluations using age-appropriate instruments provided in the protocol.
8. Had been informed of the nature of the study and informed consent and assent (as appropriate) have been obtained from the legally responsible parent(s)/legal guardian(s) and subject, respectively, in accordance with IRB requirements.

   To participate in the PK Period, subjects had:
9. Been hospital inpatients, expected to be hospitalized for up to 72 hours following the initial administration of oxymorphone ER.
10. An indwelling access catheter in place for blood sampling.

Exclusion Criteria:

1. Had known allergies or sensitivities to oxymorphone or other opioid analgesics.
2. Had a known sensitivity to any component of the oxymorphone ER.
3. Had a life expectancy <3 months.
4. Was pregnant and/or lactating.
5. Had cyanotic heart disease.
6. Had respiratory, hepatic, renal, neurological, psychological disease, or any other clinically significant condition that would, in the Investigator's opinion, preclude participation in the study.
7. Had abdominal trauma that would interfere with absorption of oxymorphone ER.
8. Had increased intracranial pressure.
9. Had a respiratory condition requiring intubation.
10. Had a history of uncontrolled seizures that were not managed with anticonvulsants.
11. Had prior history of substance abuse or alcohol abuse.
12. Had taken a monoamine oxidase inhibitor (MAOI) within 14 days prior to the start of oxymorphone ER.
13. Had taken oxycodone or oxymorphone within 48 hours prior to Baseline.
14. The investigator anticipated that the subject and/or parent(s)/legal guardian(s) was unable to comply with the protocol.
15. The subject (and/or parent[s]/legal guardian[s]) was (were) unable to communicate effectively with study personnel.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2013-03-11 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Score using FPS-R | 14 Days Post Last Dose
  Faces Pain Scale - Revised (FPS-R) self-report measure used to assess pain intensity in participants ages 7 - ≤12 years old, consists of 6 faces, visually representing increasing changes in pain intensity bounded on the left by "no pain" and on the right by "very much pain".
Pain Intensity Score using NRS-11 | 14 Days Post Last Dose
  Numerical Rating Scale (NRS-11) is an 11-point categorical numerical rating scale to assess pain intensity in participants ages 13 - ≤17 years old. The scale is anchored on the left with "No Pain" and is anchored on the right with "Worst Possible Pain".

CONTACTS AND LOCATIONS:
Overall Officials: Saji Vijayan, Study Director — Endo Pharmaceuticals
Locations (5):
- United States (5):
  - Endo Clinical Trial Site #3, Orange, California
  - Endo Clinical Trial Site #5, New Orleans, Louisiana
  - Endo Clinical Trial Site #1, Oklahoma City, Oklahoma
  - Endo Clinical Trial Site #4, Pittsburgh, Pennsylvania
  - Endo Clinical Trial Site #2, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP